CLINICAL TRIAL: NCT04155593
Title: In-office Assessment of Voiding Function Following Botox Injection for Overactive Bladder; Does Measuring Post Void Residual Impact Management
Brief Title: In-office Assessment of Voiding Function Following Botox Injection for Overactive Bladder
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 19-091
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-11

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to describe the rates of elevated post void residual (PVR) (defined as >200mL) in Cincinnati Urogynecology Associates patients following Botox injection, as well as to document how many patients required treatment with clean intermittent self-catheterization (CISC).

DETAILED DESCRIPTION:
Approximately 16% of all women have symptoms of overactive bladder (OAB), whereas 30% of the elderly population are affected. Patients who do not respond to, or cannot tolerate, first and second line therapy with behavioral modifications and pharmacotherapy are offered additional treatment options. Third line therapy involves injection of onabotulinumtoxinA (Botox©, Allergen) into the bladder detrusor muscle.

Botox was approved for use for the diagnosis of OAB in 2013. Cincinnati Urogynecology Associates (CUA), TriHealth Inc. has incorporated intravesical Botox injections into the management algorithm for refractory OAB, since 2014. Currently, patients who fail to improve after a trial of first and second line therapy are offered treatment with Botox.

The standard practice is to request patients return to the office for a routine PVR measurement using straight catheterization within approximately two-four weeks following their Botox injection. This is done regardless if patients are exhibiting symptoms of urinary retention. Patients with an elevated PVR are treated with CISC if they are symptomatic.

Nevertheless, many studies suggest that patients are accurately able to self-identify symptoms of urinary retention, and treating asymptomatic urinary retention may not be necessary.

The investigators aim to describe how many patients with PVR >200mL had symptoms following intravesical injection of Botox for OAB.

ELIGIBILITY:
Inclusion Criteria:

* OnabotulinumtoxinA injections in the bladder for overactive bladder
* Completed a post injection appointment at which time PVR was collected (approximately 10 to 28 days following Botox injection)
* Age >18
* English speaking

Exclusion Criteria:

* OnabotulinumtoxinA injection for any other cause than overactive bladder
* Patients requiring self-catheterization at baseline
* Failure to complete a postoperative appointment within 4 weeks of Botox injection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent onabotulinumtoxinA injections for overactive bladder by one of four fellowship trained female pelvic medicine and reconstructive surgeons at TriHealth between October 1, 2015 and October 1, 2019. These patients will be identified by CPT codes recorded in the EPIC electronic medical record.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects having elevated PVR | approximately 10 to 28 days following Botox injection
  Number of subjects with PVR > 200mL following Botox injection for OAB

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Pauls, MD, Principal Investigator — TriHealth - Cincinnati Urogynecology Associates
Locations (1):
- Cincinnati Urogynecology Associates, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Aldrich ER, Pauls RN. Routine Office Assessment After OnabotulinumtoxinA Injection for Overactive Bladder Is Unnecessary to Detect Clinically Significant Voiding Dysfunction. Female Pelvic Med Reconstr Surg. 2021 Apr 1;27(4):225-229. doi: 10.1097/SPV.0000000000001001. PMID 33770805